CLINICAL TRIAL: NCT04458480
Title: Effect of Fast Inpatient Rehabilitation After Total Knee Arthroplasty
Brief Title: Effect of Fast Inpatient Rehabilitation After TKA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019113
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Total Knee Arthroplasty; Rehabilitation
Keywords: Fast Rehabilitation; Inpatient Rehabilitation; Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Group: Both exposed group and control group are undertaken TKA surgery and routine postoperative management for 2 days in orthopedics department. Exposed group patients are transferred from orthopedics department to rehabilitation department on 2nd day after TKA, and accept fast inpatient rehabilitation for 1 week before hospital discharge, while control group patients continue to accept routine peri-operative management and conventional oral instructions of exercises in orthopedics department until hospital discharge.
  Interventions: Combination Product: Fast Inpatient Rehabilitation
- Control Group: Both exposed group and control group are undertaken TKA surgery and routine postoperative management for 2 days in orthopedics department. Exposed group patients are transferred from orthopedics department to rehabilitation department on 2nd day after TKA, and accept fast inpatient rehabilitation for 1 week before hospital discharge, while control group patients continue to accept routine peri-operative management and conventional oral instructions of exercises in orthopedics department until hospital discharge.

INTERVENTIONS:
Combination Product: Fast Inpatient Rehabilitation — Routine inpatient rehabilitation protocol, administered by licensed Physical Therapist, duration period of 1.5h-2h each time, 2 times for weekdays and 1 time for weekends, totally lasting for 1 week, are applied to the exposed group. After the fast inpatient rehabilitation for 1 week, the patients can get discharged if reaching to the rehabilitation goals of symptoms of pain and swell reduced, knee flexion ≥ 90° and knee extension ≥ 0°, quadriceps femurs and hamstrings muscle strength enhanced, recovery to aided standing and walking, and acquiring of rehabilitation training methods.
  Groups: Exposed Group

SUMMARY:
Rehabilitation is an important part of the post-operative treatment after TKA by consensus. This study intends to analysis whether fast inpatient rehabilitation after TKA can improve knee joint or general function, and ultimately explore for effects and values of fast inpatient rehabilitation after TKA.

DETAILED DESCRIPTION:
Rehabilitation, which is an important part of the post-operative treatment after TKA, could effectively alleviate symptoms of pain and swell, as well as improve knee joint and general function. It has reached a consensus that post-TKA rehabilitation should contain muscle strengthening, ROM, proprioceptive, balance training and physical factor therapy, etc. This study intends to use observational cohort study methods with exposure factor of fast inpatient rehabilitation after TKA, establish a TKA exposure group and a control group of TKA without inpatient rehabilitation, analysis whether fast inpatient rehabilitation after TKA can improve knee joint or general function, and ultimately explore for effects and values of fast inpatient rehabilitation after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Initial unilateral TKA patients due to osteoarthritis, rheumatoid arthritis, etc.
* Satisfactory operative knee joint ROM: knee flexion ≥120° and extension ≥ 0°.
* Prior informed consent by patients.

Exclusion Criteria:

* Complication of other medical conditions and disability to cooperate with rehabilitation.
* Complication of other conditions affecting bilateral lower limbs such as fracture, tumor, neurologic disorder, etc.
* Deep venous thrombosis of lower limbs with exception of inter-muscular venous thrombosis.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: He/She is admitted to orthopedics department of Peking University Third Hospital and undertaken initial unilateral TKA due to osteoarthritis, rheumatoid arthritis, etc.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-07 (Actual); Primary Completion 2020-09-06 (Estimated); Study Completion 2021-03-06 (Estimated)

PRIMARY OUTCOMES:
bilateral knee Rang Of Motion (ROM) | 1 day after TKA
  bilateral knee flexion and extension ROM are measured by articular protractor
bilateral quadriceps femurs | 1 day after TKA
  measured by manual muscle test (MMT)
hamstrings muscle strength | 1 day after TKA
  measured by manual muscle test (MMT)
Hospital for Special Surgery-Knee Rating scale (HSSKR) | 1 day after TKA
  to measure knee function, with the minimum 0 and maximum 100, higher score means a better outcome
modified Barthel Index (mBI) | 1 day after TKA
  to measure ADL, with the minimum 0 and maximum 100, higher score means a better outcome
Numerical Rating Scale (NRS) for pain | 1 day after TKA
  the minimum is 0 and maximum 10, higher score means a worse outcome
NRS for pain | 6 weeks after TKA
NRS for pain | 3 months after TKA
NRS for pain | 6 months after TKA
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 day after TKA
  to measure knee function and global function, with the minimum 0 and maximum 100, higher score means a better outcome
KOOS | 6 weeks after TKA
KOOS | 3 months after TKA
KOOS | 6 months after TKA

CONTACTS AND LOCATIONS:
Overall Officials: Mouwang Zhou, MM, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes